CLINICAL TRIAL: NCT05233995
Title: Clinical Trial Phase III to Evaluate the Effectiveness of the Open Abdomen as a Bridge Therapy to Perform Transit Reconstruction in Patients With Anastomosis Dehiscence.
Brief Title: Open Abdomen and Delayed Anastomosis After Anastomotic Dehiscences to Avoid Stomas
Acronym: STOP-STOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP STOMA
Record Dates: First submitted 2021-11-19; First posted 2022-02-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Anastomotic Complication; Anastomotic Leak Small Intestine; Anastomotic Leak Large Intestine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The patients included in the experimental group will be operated on, performing the resection of the intestinal segment affected by the dehiscence, the sectioned intestinal ends will be left without anastomosis, and open abdomen therapy will be established. After surgery, the patient will be cared for in the intensive care unit where intensive resuscitation will be carried out in order to improve the general conditions of the patient. After 48 ± 24 hours, a second surgical procedure will be performed where local conditions will be evaluated and the possibility of performing a delayed anastomosis will be evaluated.
  Interventions: Procedure: Damage Control Surgery
- Control group (Active Comparator): The patients included in the control group will be operated on with a resection of the affected intestinal segment and a stoma with or without associated mucosal fistula will be performed at the same surgical time. After the procedure, the patient will be cared for in the intensive care unit in order to improve the general conditions of the patient.
  Interventions: Procedure: Damage Control Surgery

INTERVENTIONS:
Procedure: Damage Control Surgery — Delayed anastomosis

SUMMARY:
Phase III clinical trial to evaluate the efficacy of the open abdomen as bridging therapy to perform transit reconstruction in patients with anastomotic dehiscence. It is a randomized controlled single-center study that will be carried out at the Virgen del Rocío University Hospital in Seville.

DETAILED DESCRIPTION:
The selected patients will be those patients reoperated for an anastomotic dehiscence (intestinal, ileocolic, colo-colic or colorectal anastomosis) with localized or generalized peritonitis. Those patients with anastomosis in the middle or lower rectum will be excluded. Once selected, if all the inclusion criteria and none of the exclusion criteria are met, the patient (or family members in case the patient does not have a sufficient level of consciousness to understand and accept the information) will be informed in detail of the therapeutic options included in the study as well as their randomization and will sign the informed consent, understanding and accepting all the information.

The patients included in the experimental group will be operated on, performing the resection of the intestinal segment affected by the dehiscence, the sectioned intestinal ends will be left inside the abdomen without anastomosis, and open abdomen with Vacuum Assisted Closure therapy will be established. After surgery, the patient will be cared for in the intensive care unit where resuscitation will be carried out in order to improve the patient's general conditions. After 48 ± 24 hours, a second surgical procedure will be carried out where local conditions will be evaluated in order to decide performing a delayed anastomosis.

The patients included in the control group will be operated on with the resection of affected intestinal segment and a stoma with or without associated mucosal fistula will be performed at the same surgical time. After the procedure, the patient will be cared for in the intensive care unit in order to improve the general conditions of the patient.

The main efficacy variable will be the stoma generation during each of the interventions and the main safety variable will be mortality in both groups. Other secondary variables will be collected, such as: Intensive Care Unit (ICU) stay, need for a non planned re-intervention, early and late complications related to surgery, complications associated with the use of an open abdomen technique.

A descriptive analysis of the quantitative variables will be carried out using the size, means and standard or median deviations and percentiles, the bilateral 95% confidence interval and range (minimum and maximum) or P50 [P25 - P75].

The relationship between dichotomous qualitative variables will be studied using the chi-square test, or Fisher's exact statistic if necessary. The effect of each of the treatment groups on the outcome variables will be measured by calculating the relative risk (RR) together with its 95% confidence interval (CI).

In all patients, a follow-up visit will be carried out at one month, at 6 months and at 12 months after surgery in order to evaluate the associated complications and record possible adverse events.

The study will be reviewed and approved by the Seville Provincial Research and Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intestinal, ileocolic, colo-colic and colorectal anastomosis dehiscence.

Exclusion Criteria:

* Dehiscence of colorectal anastomosis in the middle or lower rectum.
* Dehiscence of esophagus-gastric or gastro-intestinal anastomosis.
* Dehiscence of a colorectal anastomosis in which it is impossible to close the rectal stump.
* Failure to sign the informed consent.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Stoma after discharge | up to 57 months
  To assess the efficacy of the open abdomen surgical strategy with delayed anastomosis in patients requiring reoperation for anastomotic dehiscence. Number of stoma after discharge

SECONDARY OUTCOMES:
Mortality | up to 57 months
  To assess the mortality rate in each treatment group.
Intensive Care Unit stay | up to 57 months
  To measure the stay in the ICU of the patients in the experimental group and the control group
Complications of open abdomen | up to 57 months
  To identify the complications associated with the use of open abdomen therapy.
Early complications | up to 57 months
  To evaluate early complications in both groups.
Late complications | up to 57 months
  To collect the late complications associated with each of the therapeutic options.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Durán Muñoz-Cruzado, PhD, Principal Investigator — Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Locations (1):
- Hospital Universitario Virgen del Rocío, Sevilla, Seville, Spain